CLINICAL TRIAL: NCT03801642
Title: Randomized Controlled Pilot Trial Of Dapagliflozin In Alzheimer's Disease
Brief Title: Dapagliflozin In Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jeff Burns, MD (Other)
Responsible Party: Sponsor-Investigator, Jeff Burns, MD, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dapa in AD
Record Dates: First submitted 2018-12-21; First posted 2019-01-11 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): 10 mg dapagliflozin oral tablet taken once daily for 12 weeks
  Interventions: Drug: Dapagliflozin
- Matching placebo (Placebo Comparator): Placebo oral tablet taken once daily for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg oral tablets taken once daily for 12 weeks
  Other Names: Farxiga
  Arms: Dapagliflozin
Other: Placebo — Placebo tablet (matched in size and color to active tablet) taken once daily for 12 weeks
  Arms: Matching placebo

SUMMARY:
This is a pilot randomized controlled trial in individuals with probable Alzheimer's disease testing the effects of 10 mg dapagliflozin, taken daily for 12 weeks, on cerebral n-acetyl aspartate (NAA) levels using magnetic resonance spectroscopy (MRS). The investigators will also examine the safety and tolerability of dapagliflozin and explore the effects on systemic NAA levels in blood and urine, cerebral metabolism (fluorodeoxyglucose [FDG] PET), systemic metabolic biomarkers that indicate and quantify secondary metabolic effects, and cognitive performance.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, parallel group, 12-week study performed at a single site (University of Kansas Alzheimer's Disease Center) to investigate the effect of dapagliflozin in participants with probable AD (MMSE 15-26 inclusive). A total of 48 participants will be enrolled with 2:1 randomization to 10mg dapagliflozin once daily (n=32) for 12 weeks vs matching placebo (n=16).

The primary objective of the study is to assess the effect of 12 weeks of 10mg dapagliflozin once daily on cerebral NAA (a proxy measure of mitochondrial mass) in participants with AD.

Procedures will include phlebotomy, urine collection, MRI/MRS, FDG-PET, cognitive testing, DEXA scanning, and indirect calorimetry at baseline and 12 weeks to assess these outcomes:

* N Acetyl-Aspartate (NAA): Cerebral NAA (as measured by MRS) and Systemic NAA levels (in blood and urine)
* Cerebral metabolism (by FDG PET)
* Systemic metabolic effects: Lipids (total cholesterol, LDL, HDL), Plasma beta-hydroxybutyrate, Insulin resistance (Hemoglobin A1c, glucose and insulin during tolerance testing), Catabolic/Anabolic state [activated AKT and MTOR], Mitochondrial function measures [platelet cytochrome oxidase and citrate synthase], Inflammatory mechanisms [MCP-1, eotaxin, TNF alpha, CRP], Body composition (DEXA scanning for fat and lean mass), Resting metabolic rate (indirect calorimetry),
* Cognitive effects will be assessed at baseline and week 12 using the Alzheimer's Disease Assessment Scale-Cognitive Subscale 14 (ADAS-Cog14) and individual tests of Logical Memory I and II, Trailmaking A and B, and Stroop Word Color Test.
* 12 participants will be enrolled in an optional MRI/MRS sub-study with repeat MRI/MRS prior to randomization to assess scan-rescan reliability of the NAA measure.

Safety and tolerability of dapagliflozin (10mg daily) will be monitored throughout the study and formally at every study visit to assess the incidence and severity of AEs and the rate of discontinuations due to AEs. Safety assessments will include measuring vital signs and body weight, safety labs (including a comprehensive metabolic panel [CMP] and complete blood count [CBC] with differential) and physical and neurological examinations at screening and at end of treatment (EOT).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Have a diagnosis of probable AD per McKhann et al. criteria
3. Have a body mass index (BMI) ≥23
4. Age 50-85
5. Have a Mini Mental Status Exam (MMSE) score of 15-26 (inclusive) at screening visit
6. Have a reliable and competent study partner who is willing to accompany the participant to all study visits, monitor compliance of study medication administration, and observe/report any changes in the participant's health throughout the study duration
7. Are on stable doses of concurrent medications for at least 4 weeks prior to the screening visit
8. Speaks English as his/her primary language.
9. Females of child-bearing potential (i.e., pre-menopausal) must have a negative urine pregnancy test at the screening visit and must agree to use of contraception throughout the trial and for 30 days after the last dose of study medication. The approved methods of contraception are abstinence, the consistent use of an approved oral contraceptive (birth control pill or "the pill"), an intrauterine device (IUD), hormonal implants, contraceptive injection, double barrier method (diaphragm with spermicidal gel or condom with contraceptive foam).

Exclusion Criteria:

1. Received an investigational product in another clinical study during the last 4 weeks prior to screening
2. Diagnosis of Type 1 diabetes
3. Diagnosis of Type 2 diabetes treated with insulin, sulfonylureas, glucagon like peptide1 receptor agonists (GLP-1), thiazolidinedione (TZD) or SGLT2 inhibitors (metformin monotherapy is allowed).
4. Estimated Glomerular Filtration Rate (eGFR; MDRD) <45 mL/min at screening or unstable renal disease.
5. Any condition when MRI is contraindicated such as, but not limited to, having a pacemaker or claustrophobia.
6. Severe hepatic injury and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN. Total bilirubin >2.0 mg/dL (34.2 μmol/L)
7. Intolerance or allergy to dapaglifozin or any other SGLT2 inhibitor or any other substance in the tablets.
8. Dementia due to causes other than AD
9. History of recurrent urinary tract infection
10. Active mycotic genital infection
11. History of bladder cancer
12. History of diabetic ketoacidosis
13. Potentially confounding, serious, or unstable medical conditions such as:

    1. cancer within the past 3 years (except basal cell, squamous cell, or localized prostate cancer)
    2. a recent cardiac event (i.e. heart attack, angioplasty, etc. within the 3 months prior to screening visit)
    3. other conditions that pose a potential safety risk or confounding factor in the investigator's opinion
14. Any abnormal physical examination assessment or vital sign assessment at the screening visit that is deemed to be clinically significant by the principal investigator.
15. Any abnormal clinical laboratory test result at the screening visit that is deemed to be clinically significant by the principal investigator.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Burns, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin | Matching Placebo
Started | 30 | 16
Completed | 30 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Matching Placebo | Total
Number analyzed (Participants) | 30 | 16 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (7.9) | 71.8 (8.1) | 71.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 18 | 12 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 24 | 13 | 37
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 28 | 16 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Cerebral N Acetyl-Aspartate (NAA) / Cerebral Creatine
Description: Estimated mean change from baseline in the ratio of cerebral NAA/ cerebral Creatine as measured by MRI Spectroscopy.
Time Frame: 12 weeks
Population: All participants completing MRI spectroscopy at baseline and week-12, where data for both scans passed the data quality criteria.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Dapagliflozin | Matching Placebo
Number analyzed (Participants) | 28 | 15
Ratio | 1.49 (0.11) | 1.42 (0.09)

2. Other Pre Specified Outcome: Systemic NAA Levels
Description: NAA concentration levels in blood and urine using UPLC-MS/MS method
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Other Pre Specified Outcome: FDG PET Metabolism (Standard Uptake Value Ratio)
Description: FDG PET measures reflecting cerebral metabolism standardized to the uptake value of the cerebellum and standardized uptake value ratios (SUVR) will be calculated from native-space ROIs.
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Total Cholesterol
Description: Total cholesterol level
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: LDL Cholesterol
Description: LDL cholesterol level
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: HDL Cholesterol
Description: HDL cholesterol level
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Plasma Beta-hydroxybutyrate
Description: Plasma beta-hydroxybuteryate levels (ketones)
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Hemoglobin A1C
Description: Hemoglobin A1C
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Glucose Area Under the Curve
Description: Glucose area under the curve will be calculated based on glucose levels during a 120 minute oral glucose tolerance test.
Time Frame: 12 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Insulin Area Under the Curve
Description: Insulin area under the curve will be calculated based on insulin levels during a 120 minute oral glucose tolerance test.
Time Frame: 12 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Activated AKT Levels
Description: Activated AKT will be measured in lymphocytes immunochemically.
Time Frame: 12 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: MTOR Phosphorylation
Description: MTOR phosphorylation will be measured in lymphocytes
Time Frame: 12 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Platelet Cytochrome Oxidase Activity
Description: Cytochrome Oxidase Vmax activity is determined as a pseudo first order-rate constant (sec-1/mg protein) by measuring the oxidation of reduced cytochrome c at 550 nm
Time Frame: 12 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Monocyte Chemotactic Protein 1 (MCP-1)
Description: MCP-1, a measure of inflammation, will be measured in platelet free plasma using ELISA.
Time Frame: 12 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Eotaxin-1
Description: Eotaxin-1, a measure of inflammation, will be measured in platelet free plasma using ELISA.
Time Frame: 12 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Tumor Necrosis Factor (TNF) - Alpha
Description: TNF-alpha, a measure of inflammation, will be measured in platelet free plasma using ELISA.
Time Frame: 12 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: C-Reactive Protein (CRP)
Description: CRP, a measure of inflammation, will be measured in platelet free plasma using ELISA.
Time Frame: 12 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Total Fat Mass
Description: Body composition will be assessed using dual energy x-ray absorptiometry (GE Lunar iDEXA) to determine fat-free mass, fat mass, and percent body fat at baseline, and week 12
Time Frame: 12 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Total Lean Mass
Description: as for outcome 18
Time Frame: 12 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Resting Metabolic Rate
Description: Resting metabolic rate will be assessed using indirect calorimetry which measures CO2 production and O2 consumption to calculate total energy produced.
Time Frame: 12 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: ADAS-Cog 14
Description: Cognitive performance as measured by total score on the ADAS-cog 14.
Time Frame: 12 weeks
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Trailmaking B
Description: Cognitive performance as measured by Trailmaking B
Time Frame: 12 weeks
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Stroop Word Color Test
Description: Cognitive performance on the Stroop Word Color test.
Time Frame: 12 weeks
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Logical Memory II
Description: Memory performance as measured by the Logical Memory II test.
Time Frame: 12 weeks
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Number of Adverse Events
Description: Total number of adverse events considered related to the study medication
Time Frame: 14 weeks
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Number of Discontinuations Due to Adverse Events
Description: Number of participants who stop taking the study medication due to adverse events
Time Frame: 14 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data was collected from week 0 to week 12
Description: Does not differ
Arm/Group | Dapagliflozin | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/16
Other Adverse Events (participants affected / at risk) | 13/30 | 8/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=30) | Matching Placebo (N=16)
Cold (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Basal Cell Carcinoma Removal (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Discomfort with Urination (Renal and urinary disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dizziness (Ear and labyrinth disorders) | 4 (4) | 0 (0)
Increase in Frequency of Urination (Renal and urinary disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatigue (Endocrine disorders) | 1 (1) | 1 (1)
Poison Ivy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hornet Sting (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Worsening in Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Upper Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upset Stomach (Gastrointestinal disorders) | 0 (0) | 1 (1)
Right Big Toe Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT03801642/Prot_SAP_000.pdf